CLINICAL TRIAL: NCT02430428
Title: Use of the VisuMax™ Femtosecond Laser Lenticule Removal Procedure for the Correction of Myopia Wtih or Without Astigmatism
Brief Title: Correction of Myopia Wtih or Without Astigmatism Using the VisuMax™ Femtosecond Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carl Zeiss Meditec, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VisuMax-2014-1
Record Dates: First submitted 2015-04-23; First posted 2015-04-30 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Myopia; Astigmatism
MeSH Terms: conditions — Myopia; Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VisuMax lenticule removal (Experimental): VisuMax femtosecond laser sphere-only or spherocylindrical treatment
  Interventions: Device: Carl Zeiss Meditec VisuMax Femtosecond Laser

INTERVENTIONS:
Device: Carl Zeiss Meditec VisuMax Femtosecond Laser — VisuMax femtosecond laser sphere-only or spherocylindrical treatment

SUMMARY:
The objective of this clinical trial is to evaluate the safety and effectiveness of the Carl Zeiss Meditec VisuMax™ Femtosecond Laser lenticule removal procedure for the reduction or elimination of myopia from ≥ -1.00 D to ≤ -10.00 D with ≤ -3.00 D cylinder (myopia with or without astigmatism) and MRSE ≤ -11.50 D.

DETAILED DESCRIPTION:
This is a prospective multi-center clinical trial in which a maximum of 360 eyes of 360 consecutive subjects will be enrolled and treated with the VisuMax™ Femtosecond Laser. The study will be conducted at up to 8 clinical sites.

Subjects will be screened for eligibility, and informed consent will be obtained from those who meet screening criteria and are interested in participating in the study. Eligible subjects will be examined preoperatively to obtain a medical history and to establish a baseline ocular condition. Baseline and postoperative measurements will include manifest refraction, cycloplegic refraction, distance visual acuity (best corrected and uncorrected), slit-lamp examination, fundus examination, corneal topography, central corneal pachymetry, mesopic pupil measurement, wavefront analysis, mesopic contrast sensitivity, and intraocular pressure (IOP).

Only eyes with astigmatism ≥ -0.75 D to ≤ -3.00 D targeted for the full distance manifest spherocylindrical refraction, or eye(s) with astigmatism < -0.75 D targeted for the full distance manifest sphere-only refraction, will be enrolled into the study.

Subjects must have astigmatism ≤ -3.00 D in the eye to be treated. Eyes with astigmatism ≥ -0.75 D to ≤ -3.00 D will receive a spherocylindrical treatment. Eyes with astigmatism < -0.75 D will receive a sphere-only treatment.

Operative eyes with astigmatism ≥ -0.75 D to ≤ -3.00 D must be targeted for the full distance manifest spherocylindrical refraction. Operative eye(s) with astigmatism < -0.75 D must be targeted for the full distance manifest sphere-only refraction.

Monovision treatments and retreatments of the study eye will not be allowed during the course of the study. Bilateral investigational treatments will not be allowed during the study.

Safety and effectiveness criteria from the American National Standard for Ophthalmics (ANSI Z80.11-2012) - Laser Systems for Corneal Reshaping will be utilized in the evaluation of the VisuMax Femtosecond Laser.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects age 22 years of age and older;
2. Myopia from ≥ -1.00 D to ≤ -10.00 D with ≤ -3.00 D cylinder and MRSE ≤ -11.50 D in the eye to be treated;
3. A stable refraction for the past year, as demonstrated by a change in MRSE of ≤ 0.50 D in the eye to be treated;
4. A difference between cycloplegic and manifest refractions of < 0.75 D spherical equivalent in the eye to be treated;
5. UCVA worse than 20/40 in the eye to be treated;
6. BSCVA at least 20/20 in the eye to be treated;
7. Discontinue use of contact lenses for at least 2 weeks (for hard lenses) or 3 days (for soft lenses) prior to the preoperative examination, and through the day of surgery;
8. All contact lens wearers must demonstrate a stable refraction (within ±0.5 D), as determined by MRSE, on two consecutive examinations at least 1 week apart, in the eye to be treated;
9. Central corneal thickness of at least 500 microns in the eye to be treated;
10. Willing and able to return for scheduled follow-up examinations;
11. Able to provide written informed consent and follow study instructions in English

Exclusion Criteria:

1. Mesopic pupil diameter >8.0 mm;
2. Cylinder > -3.00 D;
3. Treatment depth is less than 250 microns from the corneal endothelium;
4. Eye to be treated is targeted for monovision;
5. Fellow eye has BSCVA worse than 20/40;
6. Keratometry readings via Sim-K values less than 40.00 D;
7. Abnormal corneal topographic findings, e.g. keratoconus, pellucid marginal degeneration in either eye;
8. History of or current anterior segment pathology, including cataracts in the eye to be treated;
9. Clinically significant dry eye syndrome unresolved by treatment in either eye;
10. Residual, recurrent, active ocular or uncontrolled eyelid disease, corneal scars or other corneal abnormality such as recurrent corneal erosion or severe basement membrane disease in the eye to be treated;
11. Ophthalmoscopic signs of progressive or unstable myopia or keratoconus (or keratoconus suspect) in either eye;
12. Irregular or unstable (distorted/not clear) corneal mires on central keratometry images in either eye;
13. History of ocular herpes zoster or herpes simplex keratitis;
14. Deep orbits, strong blink, anxiety, pterygium, or any other finding suggesting difficulty in achieving or maintaining suction;
15. Difficulty following directions or unable to fixate;
16. Previous intraocular or corneal surgery of any kind in the eye to be treated, including any type of surgery for either refractive or therapeutic purposes;
17. History of steroid-responsive rise in intraocular pressure, glaucoma, or preoperative IOP > 21 mmHg in either eye;
18. History of diabetes, diagnosed autoimmune disease, connective tissue disease or clinically significant atopic syndrome;
19. Immunocompromised or requires chronic systemic corticosteroids or other immunosuppresive therapy that may affect wound healing;
20. History of known sensitivity to planned study medications;
21. Participating in any other ophthalmic drug or device clinical trial during the time of this clinical investigation;
22. Pregnant, lactating, or of child-bearing potential and not practicing a medically approved method of birth control.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2015-03; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Number of subjects with MRSE within ± 1.00 D and ± 0.50 D | 1 Year
  Predictability: Decrease in manifest refraction spherical equivalent (MRSE) to within ± 1.00 D and ± 0.50 D of the intended refractive outcome at the point at which stability is first reached
Improvement in UCVA following treatment | 1 Year
  The uncorrected visual acuity of 20/40 or better for eyes targeted for emmetropia at the postoperative interval at which stability has been established
Preservation of Best-Spectacle Corrected Visual Acuity (BSCVA) | 1 Year
  Preservation of Best-Spectacle Corrected Visual Acuity (BSCVA):
  1. In eyes with preoperative BSCVA 20/20 or better, the percentage of eyes with BSCVA worse than 20/40 at the postoperative interval at which stability has been established
  2. The percentage of eyes with BCVA loss ≥ 2 lines
Number of subjects with induced MRCyl > 2.00 D | 1 Year
  Induced manifest refractive astigmatism: The percentage of eyes treated for spherical myopia only with induced manifest refractive cylinder of > 2.00 D at the postoperative interval at which stability has been established
Incidence of Adverse Events | 1 Year
  Incidence of Adverse Events: The rate of each type of adverse event will be summarized
Change in Contrast Sensitivity | 1 Year
  Contrast Sensitivity: Mean of "within-eye" loss of contrast sensitivity from baseline to 12 months will be provided with the 1-sided 95% confidence interval for each spatial frequency. Percentage of eyes showing ≥ 0.3 log units loss at two or more spatial frequencies at the last available postoperative visit will be calculated.

SECONDARY OUTCOMES:
Patient Symptoms | 1 Year
  Patient Symptoms: Will be considered as a secondary safety variable and will be evaluated via a subject questionnaire.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Dishler Laser Institute, Greenwood Village, Colorado
  - Discover Vision Centers, Leawood, Kansas
  - Vance Thompson Vision, Sioux Falls, South Dakota
  - Slade and Baker Vision Center, Houston, Texas
  - Davis Duehr Dean, Madison, Wisconsin